CLINICAL TRIAL: NCT02048696
Title: Effect of Exercise Training on Left Ventricular Function in Patients Post Myocardial Infarction: The EXercise Interval Training - V Study
Brief Title: Effect of Exercise Training on Left Ventricular Function in Patients Post Myocardial Infarction
Acronym: EXIT-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13-1509
Record Dates: First submitted 2014-01-22; First posted 2014-01-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Myocardial Infarction; Heart Failure; Coronary Artery Disease
Keywords: Exercise training; High intensity interval training; left ventricular systolic function; G-protein related kinase 2; heart failure; myocardial infarction; coronary artery disease; beta adrenergic receptor
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Coronary Artery Disease | interventions — Secondary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): Secondary prevention and cardiac rehabilitation clinic of the Montreal Heart Institute. Subjects will undergo twice weekly exercise training with high intensity interval training for a period of 12 weeks.
  Interventions: Other: Secondary prevention and cardiac rehabilitation clinic
- control (No Intervention): Individuals in this group are offered current ACC/AHA recommendations on physical activity in patients post-myocardial infarction.

INTERVENTIONS:
Other: Secondary prevention and cardiac rehabilitation clinic — Secondary prevention and cardiac rehabilitation clinic of the Montreal Heart Institute. Subjects will undergo twice weekly exercise training with high intensity interval training for a period of 12 weeks.
  Arms: Exercise training

SUMMARY:
Patients who have suffered a heart attack are at risk of developing worsening heart function and heart failure. Exercise training has a beneficial effect on heart function and prevents heart failure. The aim of the current study is to investigate the effect of exercise training on heart function in patients who have suffered a heart attack.

DETAILED DESCRIPTION:
Patients who have suffered a myocardial infarction are at significant risk for developing heart failure and progressive left ventricular dysfunction One of the proposed mechanisms responsible for this observation is reduction in myocardial beta-adrenergic receptor density due to elevated cell membrane protein G - protein coupled receptor kinase -2 (GRK2).

It is known that exercise training preserves heart function in patients who have suffered a myocardial infarction. The mechanism for this is not clear.

The purpose of this study is to examine the effect of exercise training on myocardial function and GRK2 levels in patients who have suffered a myocardial infarction, with the hypothesis that exercise training in this population reduces GRK2 levels and preserves or improves myocardial function.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Complete revascularization: no residual major epicardial coronary artery coronary stenosis ≥ 70%; no residual left main coronary stenosis ≥ 40%.
* Stage A-C heart failure, New York Heart Association class I-III.
* Stable dose of medications during the 4 weeks prior to enrolment.
* Able to perform a maximal cardiopulmonary stress test.
* Capacity and willingness to provide sign informed consent.

Exclusion Criteria:

* Pregnant
* Coronary artery bypass surgery: patients post coronary artery bypass graft exhibit wall motion abnormalities that may interfere with speckle tracking analysis.
* Incomplete revascularization with major epicardial coronary artery (left anterior descending, circumflex, or right coronary) stenosis ≥ 70%.
* Myocardial necrosis in the absence of significant flow limiting coronary artery stenosis or thrombosis, with the exception of documented STEMI and successful thrombolytic therapy resulting on no significant residual epicardial coronary artery stenosis.
* Significant valvular disease that is greater than moderate in severity
* History of non-ischemic cardiomyopathy (dilated, restrictive, infiltrative cardiomyopathy, hypertrophic, LV non compaction, or Takotsubo cardiomyopathy)
* Significant resting ECG abnormalities that preclude accurate speckle tracking.
* Paced rhythm.
* left bundle branch block
* Atrial arrhythmias (ex. persistent/permanent atrial fibrillation, atrial flutter).
* Frequent ventricular ectopics
* Significant ventricular arrhythmias (non-sustained ventricular tachycardia or syncope).
* New York Heart Association class IIIb - IV symptoms.
* Severe LV systolic dysfunction (Ejection fraction ≤ 30%)
* Active decompensated heart failure with orthopnea or paroxysmal nocturnal dyspnea.
* Uncontrolled resting arterial hypertension > 180/110 mmHg.
* More than moderate systemic disease
* Chronic inflammation or infection.
* Any contraindication to exercise training or any condition limiting ability to partake in adequate exercise stress testing or training (peripheral artery disease, articular, neurologic, or psychiatric pathology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02-01 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Lymphocyte GRK2 mRNA level | at baseline and following 12 weeks exercise training intervention
  change in lymphocyte GRK2 mRNA levels

SECONDARY OUTCOMES:
Left ventricular systolic function | at baseline and following 12 weeks exercise training intervention
  change in left ventricular systolic function
Left ventricular dimensions | at baseline and following 12 weeks exercise training intervention
  Change in left ventricular dimensions
Plasma epinephrine | at baseline and following 12 weeks exercise training intervention
  change in plasma epinephrine
heart rate variability | at baseline and following 12 weeks exercise training intervention
  change change in autonomic tone
exercise capacity (VO2max) | at baseline and following 12 weeks exercise training intervention
  Change before and after exercise training
ambulatory blood pressure | at baseline and following 12 weeks exercise training intervention
  Change in awake and 24h blood pressure
Plasma brain natriuretic peptide | at baseline and following 12 weeks exercise training intervention
  change in plasma brain naturietic peptide
Maximal cardiac output and stroke volume using electrical bioimpedance | at baseline and following 12 weeks exercise training intervention
  change in maximal cardiac output and stroke volume
lymphocyte GRK2 protein levels | at baseline and following 12 weeks exercise training intervention
  change in lymphocyte GRK2 protein levels

OTHER OUTCOMES:
Fasting glucose | at baseline and following 12 weeks exercise training intervention
  change in fasting glucose
serum lipids | at baseline and following 12 weeks exercise training intervention
  change in serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: Anil Nigam, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Centre for preventive medicine and physical activity of the Montreal Heart Institute (Centre ÉPIC), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Trachsel LD, Boidin M, Henri C, Fortier A, Lalonge J, Juneau M, Nigam A, Gayda M. Women and men with coronary heart disease respond similarly to different aerobic exercise training modalities: a pooled analysis of prospective randomized trials. Appl Physiol Nutr Metab. 2021 May;46(5):417-425. doi: 10.1139/apnm-2020-0650. Epub 2020 Oct 23. PMID 33096006
- [Derived] Trachsel LD, Nigam A, Fortier A, Lalonge J, Juneau M, Gayda M. Moderate-intensity continuous exercise is superior to high-intensity interval training in the proportion of VO2peak responders after ACS. Rev Esp Cardiol (Engl Ed). 2020 Sep;73(9):725-733. doi: 10.1016/j.rec.2019.09.013. Epub 2019 Dec 16. English, Spanish. PMID 31837947